CLINICAL TRIAL: NCT01877759
Title: Role of Bone Marrow Derived Autologous Stem Cells + Human Umbilical Cord Derived Mesenchymal Stem Cells for the Treatment of Liver Cirrhosis
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of Mesenchymal Stem Cells in Liver Cirrhosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, Co -investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSCC/BM/2013/LS/01
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Liver Cirrhosis
Keywords: Stem cell ,liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mesenchymal stem cell (Other): hUMAN MESENCHYMAL STEM CELLS
  Interventions: Biological: Mesenchymal stem cell

INTERVENTIONS:
Biological: Mesenchymal stem cell — Intravenous dose of Mesenchymal stem cell derived from human Bone Marrow & umbilical cord , IN 6 divided doses , at interval of 1 week .

SUMMARY:
Cirrhosis is caused by sustained liver damage over several years either by alcohol, viral infection (Hepatitis B, C), a toxic substance (for eg. drugs, excess copper or iron in the liver), or by blockage of biliary system such that the liver undergoes progressive scarring that slowly replaces all of normal liver cells.(LC) represents a late stage of progressive hepatic fibrosis characterized by distortion of the hepatic architecture and formation of regenerative nodules. For this condition of disease the liver transplantation is one of the only effective therapies available ,but due to lack of donors, surgical complications, rejection, and high cost are it's serious problems.

Presently stem cells are used to be a one of the treatment for the same. So our approach is to evaluate the safety and efficacy of mesenchymal stem cell in condition of liver cirrhosis .

DETAILED DESCRIPTION:
In this study, the patients with liver cirrhosis will undergo administration of human Mesenchymal stem cell MSCs intravenously for these patients.To observe the results Liver function will be monitored by serum analysis.The levels of serum alanine aminotransferase (ALT), total bilirubin (TB), prothrombin time (PT), prealbumin(PA) and albumin (ALB) will be examined at pre-transfusion, and 6th days to 1 years post-transfusion.Also the to see Improvement evaluation by MELD score ,Quality of life ,Child-Pugh score will be done .

ELIGIBILITY:
Inclusion Criteria

* 25 -65 Ages Eligible for Study
* Clinical diagnosis of liver cirrhosis
* Ability to comprehend the explained protocol and thereafter give an informed consent as well as sign the required Informed Consent Form (ICF) for the study.
* Expecting lifetime is over three years
* Ready to come all visits

Exclusion Criteria:

* History of life threatening allergic or immune-mediated reaction
* Positive test results for HIV and AIDS complex ,HCV , HbsAg and Syphilis
* Malignancies
* Sepsis
* Vital organs failure
* Pregnant or lactating women
* Subject who has been transplanted recently
* If the investigator or treating physician feels that the Subject with any disease or condition would interfere with the trial or the safety of patient

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in Liver function tests | 6 month
  1) Improvement of Liver Function tests liver functions( Albumin (ALB), Alanine aminotransferase (ALT), Aspartate Aminotransferase (AST), Prealbumin(PA), total bilirubin (TB), and direct bilirubin (DB) kidney function Blood urea nitrogen (BUN), Urea (UA), and Crea (Cr)),international normalized ratio (INR) in Liver Cirrhosis Patients

SECONDARY OUTCOMES:
Changes in liver function according to Child-Pugh | 6 MONTH
Changes in liver function according to MELD Score | 6 MONTH
Improvement in QUALITY OF LIFE SCALE (QOL) | 6 month

OTHER OUTCOMES:
Changes of any clinical symptoms like abdominal distension, appetite, debilitation | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, MS ORTHO, Principal Investigator — Chaitanya Hospital
Locations (1):
- Chaitanya Hospital, Pune, Maharashtra, India